CLINICAL TRIAL: NCT03249428
Title: Community-Based Participatory Action Pragmatic Randomized Controlled Trial Using Nicotine Mouth Spray for Tobacco Dependence in the Systemically Disadvantaged Population
Brief Title: Cytisine vs Nicotine Replacement Therapy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20240335-01H
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Tobacco Dependence; COPD Asthma; Mental Illness; Substance Use
MeSH Terms: conditions — Tobacco Use Disorder; Mental Disorders; Substance-Related Disorders | interventions — cytisine; Nicotine Replacement Therapy

STUDY DESIGN:
Intervention Model Description: 3-yr multi-centre pragmatic Randomized Controlled Trial (RCT) to compare effectiveness of nicotine e-cigarettes (e-cigs) (with counseling) with peer-led PROMPT strategy (nicotine replacement therapy (NRT) and counseling) for tobacco dependence in the inner city population.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research staff analyzing the data and members of the data and safety monitoring committee will be blinded to the treatment. allotment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nicotine Replacement Therapy (NRT) (Active Comparator): Nicotine Replacement Therapy (NRT): nicotine mouth spray, nicotine patches, nicotine gum, nicotine lozenges, and nicotine oral inhalers
  Interventions: Drug: Cytisine
- Cytisine (Active Comparator): Cytisine: 2x 1.5mg capsules 3 times a day (3mg 3 times a day).
  Interventions: Drug: Nicotine replacement therapy (NRT)

INTERVENTIONS:
Drug: Cytisine — Cytisine: 2x 1.5mg capsules 3 times a day (3mg 3 times a day).
  Arms: Nicotine Replacement Therapy (NRT)
Drug: Nicotine replacement therapy (NRT) — Nicotine Replacement Therapy (NRT): nicotine mouth sprays, nicotine patches, nicotine gum, nicotine lozenges, and nicotine oral inhalers
  Arms: Cytisine

SUMMARY:
Tobacco is the most preventable cause of disease and death in Canada. Although the tobacco use rate has substantially gone down in the general population, significant differences exist between sub-populations in Canada, for example Ottawa's highly vulnerable homeless or at-risk for homelessness population has an almost 100% tobacco smoking rate relative to 9-18% in the rest of the Canadian general population. This stark inequity in tobacco use translates into devastating healthcare outcomes such as a disproportionate amount of cancer, stroke, heart disease and death. Canadians who are homeless or at-risk for homelessness die 25 years earlier than housed Canadians, mostly due to tobacco. In order to tackle this tobacco use related inequity - a novel approach is urgently needed. Despite commonly held dogma that People Who Use Drugs (PWUD) don't want to quit smoking, many studies have demonstrated that in fact they are very interested in quitting. Moreover, the investigators pragmatic peer-led community-based action approach used in their PROMPT project has demonstrated that tobacco dependence strategies can be implemented with great success in this population. The majority of PROMPT participants reduced or quit tobacco use, in addition to reducing or quitting all other drug use. Importantly, the investigators have demonstrated that it is possible to gain the trust and engagement of marginalized populations and that researchers can create a community space that is low-threshold, safe and non-judgmental. The investigators aim to compare two tobacco dependence management strategies in the homeless (or at-risk for homelessness) multi-drug use population in Ottawa and Toronto. They will use the same peer-led approach in PROMPT with community peer researchers with lived experience; with the hope that the cost-effective community based framework derived from this trial will serve as a template for interventions and treatments in community settings for chronic diseases such as obesity and diabetes.

DETAILED DESCRIPTION:
Aim: A 3-yr multi-centre, pragmatic Randomized Controlled Trial (RCT) to compare effectiveness of Cytisine (with counseling) with peer-led PROMPT strategy (nicotine replacement therapy (NRT) and counseling) for tobacco dependence in the inner-city population.

Background: Homelessness/at-risk for homelessness populations in Canada carry disproportionate burden of many diseases, mostly due to tobacco. With smoking rates at ~100% in some subpopulations as compared to 9-18% in the general population, tobacco inequity is translated into unequal morbidity and mortality (COPD, cancers, heart diseases). Tobacco use costs the Ontario economy ~$1.6 billion/year in healthcare costs. Smoking attributable hospitalization costs ~$38.2 million/year in Ottawa alone from 2008-10. The inner-city population in Canada dies ~25 years earlier than housed Canadians, largely due to tobacco. With negligible quit rates using conventional strategies, novel approaches to address tobacco inequity are urgently needed.

Cytisine is a naturally occurring alkaloid that has long been used as a tobacco dependence treatment and management aid in Eastern Europe. Health Canada has approved Cytisine as an over-the-counter health product, and the Canadian Agency for Drugs and Technologies in Health (CADTH) has determined Cytisine to be a cost-effective tobacco dependence treatment and management aid. Given its cost-effectiveness and affordability compared to nicotine replacement therapy, Cytisine may be more accessible and effective for marginalized populations. Cytisine will be made available to study participants as a Health Canada licensed natural health product.

Study Population: 200 Toronto and Ottawa inner city homeless/at-risk for homelessness participants using poly-substances.

Primary Patient-Oriented Outcome: To assess the impact of two pragmatic tobacco dependence strategies on changes in QOL and GAINSS score measured with the EQ-5D-5L; Secondary: i) To assess effectiveness of these two strategies with biochemically validated smoking abstinence at 13 and 26 weeks; ii) To assess effectiveness of these two strategies on conventional cigarette and/or e-cigarette consumption reduction and cessation at 13 and 26 weeks; iii) To assess self-reported reduction and cessation of other substance use at 13 and 26 weeks; and; iv) To describe the safety/tolerability of Cytisine or NRT SAEs, AEs, and drop-outs due to side effects, along with therapy adherence over 26 weeks; and, v) To compare lung function using oscillometry and spirometry, as well as self-efficacy at baseline, 13 weeks, and 26 weeks; Tertiary: i) To assess the cost-effectiveness of the pragmatic tobacco dependence strategies.

Study Design: A multi-centre pragmatic RCT trial comparing Cytisine (with nicotine) with counseling or NRT with counseling for a 13-week treatment period and 26-week follow up. Similar to the real world, all participants will be given an opportunity to choose either strategy at 26 wks. The primary analysis will be change in QOL and GAINSS score measured with the EQ-5D-5L at 13 weeks between participants.

Setting: 1) The Bridge Engagement Centre, Ottawa, adjacent to the largest homeless shelter downtown; and 2) The Parkdale Activity-Recreation Centre.

Expertise: The PI is well versed in community-based research and very experienced in tobacco dependence and the target population. She led the PROMPT project, a community-based smoking cessation project engaging the same target population.

Outcomes: Pragmatic community-based participatory and peer-led research holds a tremendous potential in investigating solutions 'for the people, by and with the people'. Outcomes of this trial will aid policy makers in implementing effective programs to treat tobacco dependence in marginalized population. The cost-effective community-based framework of this trial can be used as a template for intervention in other chronic diseases (e.g. obesity or diabetes).

Timeline: The trial will require 3 yrs to complete.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Currently living in Ottawa or Toronto
* Actively used tobacco and/or nicotine products (i.e., cigarettes, vape) in the past 7 days; 2) and want to use NRT or Cytisine
* Identify as being low socioeconomic status, experiencing homelessness or at-risk for homelessness, and/or racialized
* Available for in-person follow-ups for six months

Exclusion Criteria:

* Consent declined (refusal from participant or decision maker)
* Any person who is in or planning on accessing addictions treatment (in-patient drug rehabilitation) in Ottawa or Toronto and hence will be unavailable for follow up
* Currently or recently (in the past 30 days) enrolled in any other smoking cessation program or have used/is using any e-cigs (nicotine or non-nicotine) in the past 60 days
* Terminal illness with a life expectancy of less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Overall Quality of Life | 13 weeks
  To assess impact of two tobacco dependence strategies on quality of life (QOL) measured by questionnaire (EQ-5D-5L scores)

SECONDARY OUTCOMES:
Smoking Prevalence | 26 weeks
  To assess effectiveness of two strategies (Cytisine with smoking cessation counseling vs NRT with smoking cessation counseling) with biochemically validated smoking abstinence at 13 and 26 weeks
Tobacco and e-cigarette (with nicotine) use | 26 weeks
  To assess effectiveness of these two strategies on conventional cigarette and/or e-cigarette consumption reduction and cessation at 13 and 26 weeks
Substance use | 26 weeks
  To assess self-reported reduction and cessation of other substance use at 13 and 26 weeks
Safety and tolerability of Cytisine or NRT | 26 weeks
  To describe the safety/tolerability of Cytisine or NRT SAEs, AEs, and drop-outs due to side effects, along with therapy adherence over 26 weeks
Lung function | 26 weeks
  To compare lung function using oscillometry and spirometry, as well as self-efficacy at baseline, 13 weeks, and 26 weeks

OTHER OUTCOMES:
Cost-effectiveness | 26 weeks
  To assess the cost-effectiveness of the pragmatic tobacco dependence strategies

CONTACTS AND LOCATIONS:
Overall Officials: Smita Pakhale, MD, MSc, Principal Investigator — The Ottawa Hospital, Ottawa Hospital Research Institute
Locations (1):
- The Bridge Engagement Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No